CLINICAL TRIAL: NCT01336023
Title: A 26 Week Randomised, Parallel Three-arm, Open-label, Multi-centre, Multinational Treat-to-target Trial Comparing Fixed Ratio Combination of Insulin Degludec and Liraglutide Versus Insulin Degludec or Liraglutide Alone, in Subjects With Type 2 Diabetes Treated With 1-2 Oral Anti-diabetic Drugs (OADs)With a 26 Week Extension
Brief Title: Dual Action of Liraglutide and Insulin Degludec in Type 2 Diabetes: A Trial Comparing the Efficacy and Safety of Insulin Degludec/Liraglutide, Insulin Degludec and Liraglutide in Subjects With Type 2 Diabetes
Acronym: DUAL™ I
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NN9068-3697; U1111-1119-1174 (Other: WHO); 2010-021560-15 (EudraCT Number)
Record Dates: First submitted 2011-04-13; First posted 2011-04-15 (Estimated); Results first posted 2017-06-02 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2 | interventions — IDegLira; insulin degludec; Liraglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- IDeg (Experimental)
  Interventions: Drug: insulin degludec
- IDegLira (Experimental)
  Interventions: Drug: insulin degludec/liraglutide
- Lira (Experimental)
  Interventions: Drug: liraglutide

INTERVENTIONS:
Drug: insulin degludec/liraglutide — Insulin degludec/liraglutide treatment will be initiated and titrated (individually adjusted) twice weekly according to the mean self measured plasma glucose (SMPG) (fasting). Insulin degludec/liraglutide is injected subcutaneously (under the skin) once daily.
  Arms: IDegLira
Drug: insulin degludec — Insulin degludec treatment will be initiated with 10 U and titrated (individually adjusted) twice weekly according to the mean SMPG (fasting). Insulin degludec is injected subcutaneously (under the skin) once daily.
  Arms: IDeg
Drug: liraglutide — Liraglutide will be started with 0.6 mg and subsequent 0.6 mg weekly dose escalation to 1.8 mg. Liraglutide dose of 1.8 mg/day will be continued for the remaining part of the trial. Liraglutide is injected subcutaneously (under the skin) once daily.
  Arms: Lira

SUMMARY:
This trial is conducted globally. The aim of this trial is to compare the efficacy and safety of insulin degludec/liraglutide (IDegLira) versus insulin degludec (IDeg) and liraglutide (Lira) in subjects with type 2 diabetes. Subjects are to continue their pre-trial treatment with metformin or metformin + pioglitazone throughout the entire trial.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with type 2 diabetes
* HbA1c 7.0-10.0 % (both inclusive) with the aim of a median HbA1c of 8.3%. Accordingly, when approximately 50% of the randomised subjects have a HbA1c above 8.3%, the remaining subjects randomised must have a HbA1c of below or equal to 8.3%, or when approximately 50% of the randomised subjects have a HbA1c of below or equal to 8.3%, the remaining subjects randomised must have a HbA1c above 8.3%
* Male or female, age 18 years or above (Taiwan: 20 years or above for a site 653 in Taiwan: Taichung Veterans General Hospital)
* Subjects on stable dose of 1-2 OADs (metformin [at least 1500 mg or max tolerated dose] or metformin [at least 1500 mg or max tolerated dose] + pioglitazone [at least 30 mg]) for at least 90 days prior to screening
* Body Mass Index (BMI) maximum 40 kg/m^2

Exclusion Criteria:

* Treatment with insulin (except for short-term treatment due to intercurrent illness at the discretion of the Investigator)
* Treatment with GLP-1 (glucagon-like peptide-1) receptor agonists (eg exenatide, liraglutide), sulphonylurea or dipeptidyl peptidase 4 (DPP-4) inhibitors within 90 days prior to trial
* Impaired liver function, defined as alanine aminotransferese (ALAT) at least 2.5 times Upper Normal Range (UNR) (one retest analysed at the central laboratory within a week from first sample taken is permitted with the result of the last sample being the conclusive)
* Impaired renal function defined as serum-creatinine at least 133 mcmol/l (at least 1.5 mg/dl) for males and at least 125 mcmol/l (at least 1.4) for females, or as allowed according to local contraindications for metformin (one retest analysed at the central laboratory within a week from first sample taken is permitted with the result of the last sample being the conclusive)
* Screening calcitonin at least 50 ng/L
* Subjects with personal or family history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia type 2 (MEN 2)
* Cardiac disorder defined as: congestive heart failure (NYHA class III-IV), diagnosis of unstable angina pectoris, cerebral stroke and/or myocardial infarction within the last 12 months and planned coronary, carotid or peripheral artery revascularisation procedures
* Severe uncontrolled treated or untreated hypertension (systolic blood pressure at least 180 mm Hg or diastolic blood pressure at least 100 mm Hg)
* Acute treatment required proliferative retinopathy or maculopathy (macular oedema)
* History of chronic pancreatitis or idiopathic acute pancreatitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1663 (Actual)
Dates: Start 2011-05-23 (Actual); Primary Completion 2012-05-24 (Actual); Study Completion 2012-11-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (264):
- United States (129):
  - Novo Nordisk Investigational Site, Birmingham, Alabama
  - Novo Nordisk Investigational Site, Anaheim, California
  - Novo Nordisk Investigational Site, Bermuda Dunes, California
  - Novo Nordisk Investigational Site, Concord, California
  - Novo Nordisk Investigational Site, Encino, California
  - Novo Nordisk Investigational Site, Fair Oaks, California
  - Novo Nordisk Investigational Site, Fresno, California
  - Novo Nordisk Investigational Site, Greenbrae, California
  - Novo Nordisk Investigational Site, La Jolla, California
  - Novo Nordisk Investigational Site, Long Beach, California
  - Novo Nordisk Investigational Site, Los Angeles, California
  - Novo Nordisk Investigational Site, Montclair, California
  - Novo Nordisk Investigational Site, Monterey, California
  - Novo Nordisk Investigational Site, Orange, California
  - Novo Nordisk Investigational Site, Poway, California
  - Novo Nordisk Investigational Site, San Diego, California
  - Novo Nordisk Investigational Site, San Mateo, California
  - Novo Nordisk Investigational Site, Santa Barbara, California
  - Novo Nordisk Investigational Site, Tustin, California
  - Novo Nordisk Investigational Site, Valencia, California
  - Novo Nordisk Investigational Site, Walnut Creek, California
  - Novo Nordisk Investigational Site, Colorado Springs, Colorado
  - Novo Nordisk Investigational Site, Denver, Colorado
  - Novo Nordisk Investigational Site, Golden, Colorado
  - Novo Nordisk Investigational Site, Waterbury, Connecticut
  - Novo Nordisk Investigational Site, Newark, Delaware
  - Novo Nordisk Investigational Site, Clearwater, Florida
  - Novo Nordisk Investigational Site, Delray Beach, Florida
  - Novo Nordisk Investigational Site, Fort Lauderdale, Florida
  - Novo Nordisk Investigational Site, Hialeah, Florida
  - Novo Nordisk Investigational Site, Jacksonville, Florida
  - Novo Nordisk Investigational Site, Kissimmee, Florida
  - Novo Nordisk Investigational Site, Melbourne, Florida
  - Novo Nordisk Investigational Site, Miami, Florida
  - Novo Nordisk Investigational Site, Orlando, Florida
  - Novo Nordisk Investigational Site, Pembroke Pines, Florida
  - Novo Nordisk Investigational Site, Tampa, Florida
  - Novo Nordisk Investigational Site, Atlanta, Georgia
  - Novo Nordisk Investigational Site, Columbus, Georgia
  - Novo Nordisk Investigational Site, Conyers, Georgia
  - Novo Nordisk Investigational Site, Decatur, Georgia
  - Novo Nordisk Investigational Site, Lawrenceville, Georgia
  - Novo Nordisk Investigational Site, Roswell, Georgia
  - Novo Nordisk Investigational Site, Woodstock, Georgia
  - Novo Nordisk Investigational Site, Meridian, Idaho
  - Novo Nordisk Investigational Site, Nampa, Idaho
  - Novo Nordisk Investigational Site, Avon, Illinois
  - Novo Nordisk Investigational Site, Chicago, Illinois
  - Novo Nordisk Investigational Site, Gurnee, Illinois
  - Novo Nordisk Investigational Site, O'Fallon, Illinois
  - Novo Nordisk Investigational Site, Fishers, Indiana
  - Novo Nordisk Investigational Site, Franklin, Indiana
  - Novo Nordisk Investigational Site, Indianapolis, Indiana
  - Novo Nordisk Investigational Site, Michigan City, Indiana
  - Novo Nordisk Investigational Site, Muncie, Indiana
  - Novo Nordisk Investigational Site, Crestview Hills, Kentucky
  - Novo Nordisk Investigational Site, Lexington, Kentucky
  - Novo Nordisk Investigational Site, Metairie, Louisiana
  - Novo Nordisk Investigational Site, Hyattsville, Maryland
  - Novo Nordisk Investigational Site, North East, Maryland
  - Novo Nordisk Investigational Site, Rockville, Maryland
  - Novo Nordisk Investigational Site, Buckley, Michigan
  - Novo Nordisk Investigational Site, Southfield, Michigan
  - Novo Nordisk Investigational Site, Troy, Michigan
  - Novo Nordisk Investigational Site, Chesterfield, Missouri
  - Novo Nordisk Investigational Site, Kansas City, Missouri
  - Novo Nordisk Investigational Site, Saint Charles, Missouri
  - Novo Nordisk Investigational Site, Henderson, Nevada
  - Novo Nordisk Investigational Site, Las Vegas, Nevada
  - Novo Nordisk Investigational Site, Nashua, New Hampshire
  - Novo Nordisk Investigational Site, Flemington, New Jersey
  - Novo Nordisk Investigational Site, Toms River, New Jersey
  - Novo Nordisk Investigational Site, Albany, New York
  - Novo Nordisk Investigational Site, Northport, New York
  - Novo Nordisk Investigational Site, Syracuse, New York
  - Novo Nordisk Investigational Site, The Bronx, New York
  - Novo Nordisk Investigational Site, West Seneca, New York
  - Novo Nordisk Investigational Site, Asheboro, North Carolina
  - Novo Nordisk Investigational Site, Asheville, North Carolina
  - Novo Nordisk Investigational Site, Burlington, North Carolina
  - Novo Nordisk Investigational Site, Chapel Hill, North Carolina
  - Novo Nordisk Investigational Site, Charlotte, North Carolina
  - Novo Nordisk Investigational Site, Greensboro, North Carolina
  - Novo Nordisk Investigational Site, Greenville, North Carolina
  - Novo Nordisk Investigational Site, Morehead City, North Carolina
  - Novo Nordisk Investigational Site, Shelby, North Carolina
  - Novo Nordisk Investigational Site, Statesville, North Carolina
  - Novo Nordisk Investigational Site, Winston-Salem, North Carolina
  - Novo Nordisk Investigational Site, Canton, Ohio
  - Novo Nordisk Investigational Site, Cincinnati, Ohio
  - Novo Nordisk Investigational Site, Cleveland, Ohio
  - Novo Nordisk Investigational Site, Columbus, Ohio
  - Novo Nordisk Investigational Site, Franklin, Ohio
  - Novo Nordisk Investigational Site, Kettering, Ohio
  - Novo Nordisk Investigational Site, Mason, Ohio
  - Novo Nordisk Investigational Site, Maumee, Ohio
  - Novo Nordisk Investigational Site, Oklahoma City, Oklahoma
  - Novo Nordisk Investigational Site, Beaver, Pennsylvania
  - Novo Nordisk Investigational Site, Bridgeville, Pennsylvania
  - Novo Nordisk Investigational Site, Norristown, Pennsylvania
  - Novo Nordisk Investigational Site, Philadelphia, Pennsylvania
  - Novo Nordisk Investigational Site, Pittsburgh, Pennsylvania
  - Novo Nordisk Investigational Site, East Providence, Rhode Island
  - Novo Nordisk Investigational Site, Columbia, South Carolina
  - Novo Nordisk Investigational Site, Greer, South Carolina
  - Novo Nordisk Investigational Site, Pelzer, South Carolina
  - Novo Nordisk Investigational Site, Simpsonville, South Carolina
  - Novo Nordisk Investigational Site, Spartanburg, South Carolina
  - Novo Nordisk Investigational Site, Taylors, South Carolina
  - Novo Nordisk Investigational Site, Chattanooga, Tennessee
  - Novo Nordisk Investigational Site, Kingsport, Tennessee
  - Novo Nordisk Investigational Site, Dallas, Texas
  - Novo Nordisk Investigational Site, DeSoto, Texas
  - Novo Nordisk Investigational Site, Fort Worth, Texas
  - Novo Nordisk Investigational Site, Houston, Texas
  - Novo Nordisk Investigational Site, Irving, Texas
  - Novo Nordisk Investigational Site, Killeen, Texas
  - Novo Nordisk Investigational Site, Lubbock, Texas
  - Novo Nordisk Investigational Site, San Antonio, Texas
  - Novo Nordisk Investigational Site, Sugar Land, Texas
  - Novo Nordisk Investigational Site, Ogden, Utah
  - Novo Nordisk Investigational Site, Salt Lake City, Utah
  - Novo Nordisk Investigational Site, St. George, Utah
  - Novo Nordisk Investigational Site, Burke, Virginia
  - Novo Nordisk Investigational Site, Manassas, Virginia
  - Novo Nordisk Investigational Site, Newport News, Virginia
  - Novo Nordisk Investigational Site, Virginia Beach, Virginia
  - Novo Nordisk Investigational Site, Spokane, Washington
  - Novo Nordisk Investigational Site, Milwaukee, Wisconsin
- Australia (8):
  - Novo Nordisk Investigational Site, Broadmeadow, New South Wales
  - Novo Nordisk Investigational Site, Camperdown, New South Wales
  - Novo Nordisk Investigational Site, Coffs Harbour, New South Wales
  - Novo Nordisk Investigational Site, Penrith, New South Wales
  - Novo Nordisk Investigational Site, Meadowbrook, Queensland
  - Novo Nordisk Investigational Site, Keswick, South Australia
  - Novo Nordisk Investigational Site, East Ringwood, Victoria
  - Novo Nordisk Investigational Site, Melbourne, Victoria
- Canada (13):
  - Novo Nordisk Investigational Site, Edmonton, Alberta
  - Novo Nordisk Investigational Site, Chilliwack, British Columbia
  - Novo Nordisk Investigational Site, Vancouver, British Columbia
  - Novo Nordisk Investigational Site, Winnipeg, Manitoba
  - Novo Nordisk Investigational Site, Brampton, Ontario
  - Novo Nordisk Investigational Site, Burlington, Ontario
  - Novo Nordisk Investigational Site, Cornwall, Ontario
  - Novo Nordisk Investigational Site, Hamilton, Ontario
  - Novo Nordisk Investigational Site, Mississauga, Ontario
  - Novo Nordisk Investigational Site, Toronto, Ontario
  - Novo Nordisk Investigational Site, Drummondville, Quebec
  - Novo Nordisk Investigational Site, Laval, Quebec
  - Novo Nordisk Investigational Site, Québec
- Finland (5):
  - Novo Nordisk Investigational Site, Hanko
  - Novo Nordisk Investigational Site, Helsinki
  - Novo Nordisk Investigational Site, Imatra
  - Novo Nordisk Investigational Site, Kokkola
  - Novo Nordisk Investigational Site, Oulu
- Germany (14):
  - Novo Nordisk Investigational Site, Bad Neuenahr-Ahrweiler
  - Novo Nordisk Investigational Site, Eisenach
  - Novo Nordisk Investigational Site, Esslingen am Neckar
  - Novo Nordisk Investigational Site, Frankfurt
  - Novo Nordisk Investigational Site, Grevenbroich
  - Novo Nordisk Investigational Site, Hamburg
  - Novo Nordisk Investigational Site, Herrenberg
  - Novo Nordisk Investigational Site, Hohenmölsen
  - Novo Nordisk Investigational Site, Münster
  - Novo Nordisk Investigational Site, Oldenburg
  - Novo Nordisk Investigational Site, Pohlheim
  - Novo Nordisk Investigational Site, Rehburg-Loccum
  - Novo Nordisk Investigational Site, Rehlingen-Siersburg
  - Novo Nordisk Investigational Site, Stuttgart
- Hungary (6):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Eger
  - Novo Nordisk Investigational Site, Gyula
  - Novo Nordisk Investigational Site, Pécs
  - Novo Nordisk Investigational Site, Szeged
- India (18):
  - Novo Nordisk Investigational Site, Ahmedabad, Gujarat
  - Novo Nordisk Investigational Site, Gurgaon, Haryana
  - Novo Nordisk Investigational Site, Bangalore, Karnataka
  - Novo Nordisk Investigational Site, Kochi, Kerala
  - Novo Nordisk Investigational Site, Thiruvanathapuram, Kerala
  - Novo Nordisk Investigational Site, Trivandrum, Kerala
  - Novo Nordisk Investigational Site, Indore, Madhya Pradesh
  - Novo Nordisk Investigational Site, Mumbai, Maharashtra
  - Novo Nordisk Investigational Site, Pune, Maharashtra
  - Novo Nordisk Investigational Site, Bhubaneswar, Odisha
  - Novo Nordisk Investigational Site, Jaipur, Rajasthan
  - Novo Nordisk Investigational Site, Chennai, Tamil Nadu
  - Novo Nordisk Investigational Site, Trichy, Tamil Nadu
  - Novo Nordisk Investigational Site, Kolkata, West Bengal
  - Novo Nordisk Investigational Site, Hyderabad
  - Novo Nordisk Investigational Site, Kolkata
  - Novo Nordisk Investigational Site, Patna
  - Novo Nordisk Investigational Site, Pune
- Ireland (2):
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
- Italy (8):
  - Novo Nordisk Investigational Site, Cosenza
  - Novo Nordisk Investigational Site, Forlì
  - Novo Nordisk Investigational Site, Monserrato, Cagliari
  - Novo Nordisk Investigational Site, Novara
  - Novo Nordisk Investigational Site, Olbia
  - Novo Nordisk Investigational Site, Palermo
  - Novo Nordisk Investigational Site, Siena
  - Novo Nordisk Investigational Site, Torino
- Malaysia (6):
  - Novo Nordisk Investigational Site, Cheras
  - Novo Nordisk Investigational Site, George Town
  - Novo Nordisk Investigational Site, Kota Bharu, Kelantan
  - Novo Nordisk Investigational Site, Pulau Pinang
  - Novo Nordisk Investigational Site, Putrajaya
  - Novo Nordisk Investigational Site, Seremban
- Mexico (2):
  - Novo Nordisk Investigational Site, Guadalajara, Jalisco
  - Novo Nordisk Investigational Site, Monterrey, Nuevo León
- Novo Nordisk Investigational Site, San Juan, Puerto Rico
- Russia (8):
  - Novo Nordisk Investigational Site, Kursk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Penza
  - Novo Nordisk Investigational Site, Saint Petersburg
  - Novo Nordisk Investigational Site, Saratov
  - Novo Nordisk Investigational Site, Stavropol
  - Novo Nordisk Investigational Site, Voronezh
  - Novo Nordisk Investigational Site, Vsevolozhsk
- Novo Nordisk Investigational Site, Singapore, Singapore
- Slovakia (4):
  - Novo Nordisk Investigational Site, Bratislava
  - Novo Nordisk Investigational Site, Lučenec
  - Novo Nordisk Investigational Site, Moldava nad Bodvou
  - Novo Nordisk Investigational Site, Nové Zámky
- South Africa (8):
  - Novo Nordisk Investigational Site, Port Elizabeth, Eastern Cape
  - Novo Nordisk Investigational Site, Bloemfontein, Free State
  - Novo Nordisk Investigational Site, Johannesburg, Gauteng
  - Novo Nordisk Investigational Site, Vaderbijlpark, Gauteng
  - Novo Nordisk Investigational Site, Durban, KwaZulu-Natal
  - Novo Nordisk Investigational Site, eMkhomazi, KwaZulu-Natal
  - Novo Nordisk Investigational Site, Brits, North West
  - Novo Nordisk Investigational Site, Cape Town, Western Cape
- Spain (7):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Almería
  - Novo Nordisk Investigational Site, Granada
  - Novo Nordisk Investigational Site, Partida de Bacarot
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
  - Novo Nordisk Investigational Site, Valladolid
- Taiwan (4):
  - Novo Nordisk Investigational Site, Taichung
  - Novo Nordisk Investigational Site, Tainan
  - Novo Nordisk Investigational Site, Taipei
  - Novo Nordisk Investigational Site, Taoyuan District
- Thailand (3):
  - Novo Nordisk Investigational Site, Bangkok
  - Novo Nordisk Investigational Site, Bangkoknoi, Bangkok
  - Novo Nordisk Investigational Site, Chiang Mai
- United Kingdom (17):
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Bury St Edmunds
  - Novo Nordisk Investigational Site, Carmarthen
  - Novo Nordisk Investigational Site, Dundee
  - Novo Nordisk Investigational Site, Edgbaston, Birmingham
  - Novo Nordisk Investigational Site, Fife
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Gloucester
  - Novo Nordisk Investigational Site, Headington
  - Novo Nordisk Investigational Site, Lancaster
  - Novo Nordisk Investigational Site, Letchworth Garden City
  - Novo Nordisk Investigational Site, Llantrisant
  - Novo Nordisk Investigational Site, London
  - Novo Nordisk Investigational Site, St Helens
  - Novo Nordisk Investigational Site, Stevenage
  - Novo Nordisk Investigational Site, Weston-super-Mare
  - Novo Nordisk Investigational Site, Wrexham

REFERENCES:
- [Background] Khunti K, Mohan V, Jain SM, Boesgaard TW, Begtrup K, Sethi B. Efficacy and Safety of IDegLira in Participants with Type 2 Diabetes in India Uncontrolled on Oral Antidiabetic Drugs and Basal Insulin: Data from the DUAL Clinical Trial Program. Diabetes Ther. 2017 Jun;8(3):673-682. doi: 10.1007/s13300-017-0252-9. Epub 2017 Mar 22. PMID 28332144
- [Result] Holst JJ, Buse JB, Rodbard HW, Linjawi S, Woo VC, Boesgaard TW, Kvist K, Gough SC. IDegLira Improves Both Fasting and Postprandial Glucose Control as Demonstrated Using Continuous Glucose Monitoring and a Standardized Meal Test. J Diabetes Sci Technol. 2015 Oct 6;10(2):389-97. doi: 10.1177/1932296815610124. PMID 26443290
- [Result] Vilsboll T, Vora J, Jarlov H, Kvist K, Blonde L. Type 2 Diabetes Patients Reach Target Glycemic Control Faster Using IDegLira than Either Insulin Degludec or Liraglutide Given Alone. Clin Drug Investig. 2016 Apr;36(4):293-303. doi: 10.1007/s40261-016-0376-0. PMID 26894800
- [Result] Gough SC, Bode B, Woo V, Rodbard HW, Linjawi S, Poulsen P, Damgaard LH, Buse JB; NN9068-3697 (DUAL-I) trial investigators. Efficacy and safety of a fixed-ratio combination of insulin degludec and liraglutide (IDegLira) compared with its components given alone: results of a phase 3, open-label, randomised, 26-week, treat-to-target trial in insulin-naive patients with type 2 diabetes. Lancet Diabetes Endocrinol. 2014 Nov;2(11):885-93. doi: 10.1016/S2213-8587(14)70174-3. Epub 2014 Sep 1. PMID 25190523
- [Result] Gough SC, Bode BW, Woo VC, Rodbard HW, Linjawi S, Zacho M, Reiter PD, Buse JB. One-year efficacy and safety of a fixed combination of insulin degludec and liraglutide in patients with type 2 diabetes: results of a 26-week extension to a 26-week main trial. Diabetes Obes Metab. 2015 Oct;17(10):965-73. doi: 10.1111/dom.12498. Epub 2015 Jul 1. PMID 25980900
- [Result] Kapitza C, Bode B, Ingwersen SH, Jacobsen LV, Poulsen P. Preserved pharmacokinetic exposure and distinct glycemic effects of insulin degludec and liraglutide in IDegLira, a fixed-ratio combination therapy. J Clin Pharmacol. 2015 Dec;55(12):1369-77. doi: 10.1002/jcph.549. Epub 2015 Jul 14. PMID 25998481
- [Result] King AB, Philis-Tsimikas A, Kilpatrick ES, Langbakke IH, Begtrup K, Vilsboll T. A Fixed Ratio Combination of Insulin Degludec and Liraglutide (IDegLira) Reduces Glycemic Fluctuation and Brings More Patients with Type 2 Diabetes Within Blood Glucose Target Ranges. Diabetes Technol Ther. 2017 Apr;19(4):255-264. doi: 10.1089/dia.2016.0405. Epub 2017 Mar 10. PMID 28282219
- [Result] Norwood P, Chen R, Jaeckel E, Lingvay I, Jarlov H, Lehmann L, Heller S. Rates of hypoglycaemia are lower in patients treated with insulin degludec/liraglutide (IDegLira) than with IDeg or insulin glargine, regardless of the hypoglycaemia definition used. Diabetes Obes Metab. 2017 Nov;19(11):1562-1569. doi: 10.1111/dom.12972. Epub 2017 Jul 10. PMID 28417535
- [Derived] Natale P, Green SC, Tunnicliffe DJ, Pellegrino G, Toyama T, Strippoli GF. Glucagon-like peptide 1 (GLP-1) receptor agonists for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2025 Feb 18;2(2):CD015849. doi: 10.1002/14651858.CD015849.pub2. PMID 39963952
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Countries: 19; Sites: 271; Number of sites as in parenthesis. Australia (7), Canada (14 ), Finland (5 ), Germany (12 ), Hungary (6), India (23), Ireland (2), Italy (6), Malaysia (5), Mexico (2 ), Russian Federation (11), Singapore (3), Slovakia (5), South Africa (13), Spain (8), Taiwan (3), Thailand (4), United Kingdom (16) and United States (126).
Pre-assignment Details: Subjects on metformin and/or pioglitazone treatment underwent a 26-week main trial and continued to enter an additional 26-week extension trial. Total duration of the trial was up to 55 weeks (2 weeks screening + 26 week main period + 26 week extension period + 1 week follow-up after last dose).
Groups:
- IDeg: Insulin degludec (IDeg: 100 U/mL) was injected once daily (OD) subcutaneously (s.c.) for 26 weeks (main trial) + 26 weeks (extension trial). IDeg treatment was initiated at a dose of 10 units and titrated twice weekly to the fasting glycaemic target of 4.0-5.0 mmol/L (72-90 mg/dL) based on the mean fasting self-measured plasma glucose (SMPG) from 3 preceeding measurements. Pre-trial metformin/metformin + pioglitazone treatment was continued throughout the trial.
- IDegLira: Insulin Degludec/Liraglutide (IDegLira: 100 U/3.6 mg per mL) was injected subcutaneously OD for 26 weeks(main trial) + 26 weeks (extension trial). IDegLira treatment was initiated at 10 dose steps (containing 10 units IDeg and 0.36 mg liraglutide) and titrated twice weekly to a fasting glycaemic target of 4.0-5.0 mmol/L (72-90 mg/dL) based on the mean SMPG (fasting) from 3 preceeding measurements. Pre-trial metformin/metformin + pioglitazone treatment was continued throughout the trial.
- Liraglutide: Liraglutide (6 mg/mL) was injected subcutaneously OD for 26 weeks (main trial). Liraglutide treatment was initiated at a dose of 0.6 mg/day, and subsequently increased by 0.6 mg in weekly dose escalation steps to reach maximum dose of 1.8 mg/day. Subjects continued with liraglutide 1.8 mg once daily in the 26 week extension period. Pre-trial metformin/metformin + pioglitazone treatment was continued throughout the trial.
Period: Week 0 to Week 26
Arm/Group | IDeg | IDegLira | Liraglutide
Started | 414 | 834 | 415
Exposed | 413 (1 subject withdrew before exposure to trial drug and was not included in the analysis) | 826 (8 subjects withdrew before exposure to trial drug and were not included in the analysis) | 413 (2 subjects withdrew before exposure to trial drug and were not included in the analysis)
Completed | 366 | 736 | 342
Not Completed | 48 | 98 | 73
Not completed — Adverse Event | 8 | 10 | 24
Not completed — Lack of Efficacy | 0 | 1 | 0
Not completed — Protocol Violation | 1 | 2 | 0
Not completed — Withdrawal Criteria | 34 | 69 | 40
Not completed — Unclassified | 5 | 16 | 9
Period: Week 27 to 52
Arm/Group | IDeg | IDegLira | Liraglutide
Started | 333 (From the main trial, 33 subjects were not enrolled in the extension (week 27-52).) | 665 (From the main trial, 71 subjects were not enrolled in the extension (week 27-52).) | 313 (From the main trial, 29 subjects were not enrolled in the extension (week 27-52).)
Completed | 305 | 621 | 285
Not Completed | 28 | 44 | 28
Not completed — Adverse Event | 1 | 5 | 2
Not completed — Protocol Violation | 0 | 2 | 1
Not completed — Withdrawal Criteria | 14 | 19 | 16
Not completed — Unclassified | 13 | 18 | 9

BASELINE CHARACTERISTICS:
Population: The full analysis set (FAS) included all randomised subjects and missing data was imputed using last observation carried forward (LOCF). Three subjects did not have their case book signed off due to discontinuation of an investigator's participation in the trial, hence 1 subject in each arm was excluded from the FAS.
Groups:
- Total: Total of all reporting groups
Arm/Group | IDeg | IDegLira | Liraglutide | Total
Number analyzed (Participants) | 413 | 833 | 414 | 1660
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: The number of subjects analysed in the IDeg, IDegLira and Liraglutide arms 413, 833 and 413, respectively.
  years
    number analyzed (Participants) | 413 | 833 | 413 | 1659
    (all) | 54.9 (9.7) | 55.1 (9.9) | 55.0 (10.2) | 55.0 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 213 | 398 | 206 | 817
  Male | 200 | 435 | 208 | 843
Body Weight [Mean (Standard Deviation); unit: kg] | 87.4 (19.2) | 87.2 (19.0) | 87.4 (18.0) | 87.3 (18.8)
Normalised Incremental Area under curve (AUC) [Mean (Standard Deviation); unit: mmol/L] — The area under the glucose concentration (AUC) curve during 0-4 hours after the start of a standardised meal. The incremental AUC was calculated using the trapezoidal method and the resulting area was divided length of the observation period to yield the (normalised) prandial increment in mmol/L. The data was derived from the subjects who underwent a standard meal test conducted at selected sites. Population: The number of subjects analysed in the IDeg, IDegLira and Liraglutide arms 63, 128 and 61, respectively.
  mmol/L
    number analyzed (Participants) | 63 | 128 | 61 | 252
    (all) | 4.12 (1.80) | 4.11 (2.05) | 4.12 (1.82) | 4.11 (1.93)
Glycosylated haemoglobin (HbA1c) [Mean (Standard Deviation); unit: percentage of glycosylated haemoglobin] | 8.3 (1.0) | 8.3 (0.9) | 8.3 (0.9) | 8.3 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in HbA1c (Glycosylated Haemoglobin) at Week 26.
Description: Values of mean change in HbA1c.
Time Frame: Week 0, week 26
Population: The FAS included all randomised subjects and missing data was imputed using LOCF. Three subjects did not have their case book signed off due to discontinuation of an investigator's participation in the trial; hence 1 subject from each arm was excluded from the FAS.
Measure: Mean (Standard Deviation); unit: Percentage of glycosylated haemoglobin
Arm/Group | IDeg | IDegLira | Liraglutide
Number analyzed (Participants) | 413 | 833 | 414
Percentage of glycosylated haemoglobin | -1.44 (1.03) | -1.91 (1.07) | -1.28 (1.13)
Statistical Analysis 1: Comparison: IDeg vs IDegLira; Test type: Non-Inferiority — Non-inferiority of IDegLira vs. IDeg was confirmed when 95% confidence interval for the treatment differences for change in HbA1c lies entirely below 0.3%. IDegLira minus IDeg; ANCOVA; Treatment Contrast = -0.47, 95% CI 2-sided [-0.58 to -0.36] — IDegLira minus IDeg
Statistical Analysis 2: Comparison: IDegLira vs Liraglutide; Test type: Superiority — Superiority of IDegLira over liraglutide was confirmed when the 95% confidence interval for the treatment difference for change in HbA1c lies entirely below 0%. IDegLira minus Liraglutide; ANCOVA; Treatment contrast = -0.64, 95% CI 2-sided [-0.75 to -0.53] — IDegLira minus Liraglutide

2. Secondary Outcome: Mean Change From Baseline in Body Weight at Week 26
Description: Values of mean change in body weight.
Time Frame: Week 0, Week 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | IDeg | IDegLira | Liraglutide
Number analyzed (Participants) | 413 | 833 | 414
kg | 1.6 (4.0) | -0.5 (3.5) | -3.0 (3.5)

3. Secondary Outcome: Number of Hypoglycaemic Episodes
Description: Reported hypoglycemaic episodes are number of hypoglycemic events per 100 patient years of exposure.
Time Frame: Weeks 0-26
Population: The Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparators. The missing data was imputed using LOCF. The number of subjects analysed in SAS for each arm are 412, 825 and 412, respectively.
Measure: Number; unit: Events per 100 patient years of exposure
Arm/Group | IDeg | IDegLira | Liraglutide
Number analyzed (Participants) | 412 | 825 | 412
Events per 100 patient years of exposure | 256.7 | 180.2 | 22.0

4. Secondary Outcome: Change From Baseline in Incremental Area Under the Curve 0-4h (iAUC0-4h) Derived From the Glucose Concentration Profile During Meal Test
Description: Values of mean change in normalised iAUC0-4h values based on LOCF data derived from the glucose concentration profiles during a meal test. The meal test was performed at selected sites at baseline and after 26 weeks of treatment in the main trial period. The incremental AUC was calculated using the trapezoidal method and the resulting area was divided length of the observation period to yield the (normalised) prandial increment in mmol/L using the available valid glucose observations and the associated actual elapsed time point.
Time Frame: Week 0, Week 26
Population: The number of subjects analysed were equal to study population in which the meal test was perfomed at selected sites. Missing data was imputed using LOCF.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | IDeg | IDegLira | Liraglutide
Number analyzed (Participants) | 63 | 128 | 61
mmol/L | -0.17 (1.98) | -0.87 (1.65) | -0.78 (1.62)

5. Secondary Outcome: Mean Actual Daily Insulin Dose
Description: Mean of the actual doses recorded at visit 28 (Week 26).
Time Frame: Week 26
Population: The FAS included all randomised subjects. Missing data was imputed using LOCF. For 22 subjects, the dose values were missing hence did not contribute to the analysis. The comparison was made between the insulin products IDeg and IDeglira.
Measure: Mean (Standard Deviation); unit: units
Arm/Group | IDeg | IDegLira
Number analyzed (Participants) | 408 | 816
units | 53 (28) | 38 (13)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from first day of exposure to randomised treatment of 52 weeks (26 week main period + 26 week extension period) + 7 days follow-up after the last day on randomised treatment.
Description: The Safety Analysis Set (SAS) included all subjects receiving at least one dose of the investigational product or comparators.
Arm/Group | IDeg | IDegLira | Liraglutide
Serious Adverse Events (participants affected / at risk) | 22/412 | 38/825 | 24/412
Other Adverse Events (participants affected / at risk) | 160/412 | 386/825 | 241/412
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=412) | IDegLira (N=825) | Liraglutide (N=412)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 2 (2) | 1 (1)
Angina pectoris (Cardiac disorders) | 0 (0) | 2 (2) | 2 (2)
Angina unstable (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Coronary artery dilatation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Goitre (Endocrine disorders) | 0 (0) | 0 (0) | 1 (1)
Angle closure glaucoma (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Cataract (Eye disorders) | 1 (1) | 0 (0) | 0 (0)
Necrotising retinitis (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Vitreous haemorrhage (Eye disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Biliary colic (Hepatobiliary disorders) | 0 (0) | 2 (2) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 1 (1)
Jaundice cholestatic (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abscess (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Localised infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (1)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Wrong drug administered (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Obesity (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 3 (3)
Pseudarthrosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Tendonitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer stage 0, with cancer in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Endometrial cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Inflammatory carcinoma of breast stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Pancreatic carcinoma stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Complicated migraine (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Hypertensive encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoglycaemic unconsciousness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Renal impairment (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Dysfunctional uterine bleeding (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchitis chronic (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0) | 0 (0)
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Coronary arterial stent insertion (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Coronary artery bypass (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0)
Coronary revascularisation (Surgical and medical procedures) | 1 (1) | 1 (1) | 0 (0)
Percutaneous coronary intervention (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Femoral arterial stenosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IDeg (N=412) | IDegLira (N=825) | Liraglutide (N=412)
Constipation (Gastrointestinal disorders) | 4 (4) | 26 (34) | 21 (23)
Diarrhoea (Gastrointestinal disorders) | 28 (33) | 84 (128) | 67 (94)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 28 (35) | 22 (28)
Nausea (Gastrointestinal disorders) | 16 (21) | 85 (102) | 92 (118)
Vomiting (Gastrointestinal disorders) | 10 (10) | 41 (62) | 37 (54)
Nasopharyngitis (Infections and infestations) | 52 (74) | 115 (162) | 55 (81)
Upper respiratory tract infection (Infections and infestations) | 34 (40) | 64 (79) | 33 (37)
Lipase increased (Investigations) | 18 (20) | 48 (55) | 35 (40)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 22 (23) | 30 (32)
Arthralgia (Musculoskeletal and connective tissue disorders) | 15 (23) | 30 (36) | 22 (27)
Back pain (Musculoskeletal and connective tissue disorders) | 20 (23) | 45 (45) | 23 (29)
Dizziness (Nervous system disorders) | 10 (14) | 24 (30) | 22 (25)
Headache (Nervous system disorders) | 45 (143) | 106 (207) | 60 (100)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At the end of the trial, one or more manuscripts for publication will be prepared collaboratively between Investigator(s) and Novo Nordisk. Novo Nordisk reserves the right to postpone publication and/or communication for less than 60 days to protect intellectual property.